CLINICAL TRIAL: NCT03926676
Title: One-year Clinical Assessment of Indirect Restorations Fabricated From Nano Hybrid Composite Blocks Versus Ceramic Blocks in Badly Broken Teeth (Randomized Clinical Trial)
Brief Title: Comparing Nano Hybrid Composite Blocks With Ceramic Blocks in Indirect Restorations 2. Protocol Registration:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hamsa Ashraf Abd El Menam, Hamsa Ashraf Abd El Menam, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPER-607
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: the Clinical Performance of Indirect Restoration Fabricated From Nanohybrid Cad Cam Composite Blocks and Ceramic Blocks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grandio blocks (Experimental): Nano hybrid composite blocks
  Interventions: Other: grandio blocks; Other: emax
- E max (Active Comparator): ceramic blocks
  Interventions: Other: grandio blocks; Other: emax

INTERVENTIONS:
Other: grandio blocks — nano hybrid composite blocks
Other: emax — ceramic blocks

SUMMARY:
comparing nano hybrid composite blocks grandio blocks (VOCO) with ceramic blocks (Emax) in indirect restorations using modified USPH criteria (marginal integrity) to see if there will be a significant different between two blocks

DETAILED DESCRIPTION:
Ceramic restorations are well - thought- out an excellent option to restore posterior teeth were esthetics is required and the size of the cavity preparation has surpassed the conventional for direct resin composites , Ceramic systems can syndicate esthetics with wear resistance , being considered a consistent treatment of choice ,peutzfeld evaluated , the failure rate of different restorative materials used in posterior teeth and stated that gold inlays didnt present a much lower failure rate than ceramic or composite inlays, consequently , the author suggested that other aspects besides longevity , such as esthetics , charge and number of visits should also be considered when relating treatment options

Different ceramic systems for constructing inlays and onlays restorations are available in the market, some of the ceramic restorations are made using feldspathic ceramic , the Cerec computer aided design/computer -aided manufacturing, CAD/CAM system or the hot-pressed leucite -reinforced ceramic fabricated by the conventional lost wax technique , other systems that employ alumina are available , there are three types of materials available for the dentist (glass ceramics /ceramics)resin hybrid ceramics and composite blocks Advantages of ceramic restortations are improved because of their increased translucency and light transmission ,Another advantage embraces minimal tooth reduction compared with metal ceramics , minimal thermal conductivity , they have desirable properties including their physical and mechanical properties , outstanding biocompatbility to periodontal tissues and less susceptibility to metal allergies though ceramic blocks will cause wear of opposing natural teeth ,expensive , that's why we have to shift to another material resin composite Resin composite materials have been quickly developed in the last few years , direct resin composite restorations become the gold standard for restoring intra coronal cavities , while for the extra coronal cavities , the indirect resin composite onlays be inclined to replace metallic restorations in most situations being more esthetics and conservative with lower cost.

One of the break throughs in resin composite technology is the evolution of the new resin composite blocks (Grandio blocks ) merits of grandio blocks the highest fillers content ( 86% by weight)resembles natural teeth perfectly , excellent physical values for flexural strength and abrasion , no firing required (a real one step), can be processed using any conventional milling unit , can be polished and repaired optimally , Ideal for grinding even incases with thin edges and its based on the nano hybrid technology .

ELIGIBILITY:
Inclusion Criteria:

* patients with badly broken vital teeth

good oral hygiene measures

young adults males or females

cooperative patients approving to participate in the study

Exclusion Criteria:

* patients with compromised medical history

lack of compliance

severe medical condition

severe or active periodontal disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
marginal integrity | one year
  Modified USPH criteria

CONTACTS AND LOCATIONS:
Overall Officials: shereen MO Hafez, phd, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No